CLINICAL TRIAL: NCT00624143
Title: Oral Voriconazole vs IV Low Dose Amphotericin B for Primary Antifungal Prophylaxis in Pediatric Acute Leukemia Induction:A Prospective, Randomized, Clinical Trial.
Brief Title: Antifungal Prophylaxis in Pediatric Acute Leukemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Dr. Sameer Bakhshi, Associate Professor, Medical Oncology, IRCH, AIIMS, New Delhi, Dr.Sameer Bakhshi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: antifungal prophylaxis; Dr. SAMEER BAKHSHI
Record Dates: First submitted 2008-02-19; First posted 2008-02-26 (Estimated); Last update posted 2008-02-26 (Estimated); Status verified 2008-01

CONDITIONS: Pediatric Acute Leukemia Induction
Keywords: Antifungal prophylaxis, acute leukemia induction,
MeSH Terms: interventions — Voriconazole; Amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Oral Voriconazole
  Interventions: Drug: ORAL VORICONAZOLE and IV Amphotericin B
- 2 (Active Comparator): IV Amphotericin B
  Interventions: Drug: ORAL VORICONAZOLE and IV Amphotericin B

INTERVENTIONS:
Drug: ORAL VORICONAZOLE and IV Amphotericin B — Oral Voriconazole will be given in dose of 6mg/kg 12 hourly on day1 then 4mg/kg 12 hourly daily or IV Amphotericin B 0.5 mg/kg/day weekly thrice till the completion of induction or recovery of ANC >1000/MM3 or development of fungal infection

SUMMARY:
Hypothesis:Oral Voriconazole will be as effective as intravenous Amphotericin B as antifungal prophylaxis in induction of acute leukemia (ALL, AML) in pediatric patients, with less toxicity and more convenience.

DETAILED DESCRIPTION:
RATIONALE OF STUDY:

* In induction chemotherapy for childhood acute leukemia, our experience and international studies has shown that 30% of ALL and approximately 50% of AML patients require antifungal therapy. Mortality rates associated with documented fungal infection due to opportunistic yeasts and filamentous fungi have been high, ranging from 50-90% despite use of therapeutic amphotericin B or voriconazole.
* Currently licensed drug for use in pediatric patients are amphotericin B and its lipid derivatives; 5-flucytosine; azoles like fluconazole, itraconazole, voriconazole; and caspofungin.
* Limitation with Fluconazole- inactive against Aspergilosis, C. glabrata, C. krusei, C. parapsilosis and filamentous fungi.
* Limitation with Itraconazole- erratic oral absorption of capsule form, frequent drug interactions, non availability of oral suspension form for use in very small children who would not be able to take capsules.
* Amphotericin B and Voriconazole both have proven activity against filamentous fungi and candida species.
* There is no prospective, randomised trial comparing voriconazole and amphotericin B in prophylaxis of pediatric acute leukemia during induction.

Hence there is need to study their role in prophylaxis of this infection which has a high mortality despite therapy.

Study design: Prospective, Randomized, concealed, single institutional study.

Study population:

Pediatric patients of acute leukaemia who undergo induction chemotherapy at IRCH between Jan 2008 to Dec 2009 will be eligible for the study.

Inclusion criteria:

* Patients age less than or equal to 15 years with de novo acute leukemia undergoing induction chemotherapy.
* No evidence of fungal infection at randomization
* No pneumonia at presentation.
* No systemic antifungal therapy within 7 days before randomization.

Febrile patients with no pneumonia, systemic fungal infection and hemodynamically stable will be eligible for study.

Exclusion criteria:

* Patients with baseline pneumonia.
* Laboratory evidence of significant hepatic or renal dysfunction (defined as a SGOT or SGPT more than 5 times, Total bilirubin more than 2 times and Serum creatinine more than 2 times upper limit of normal)

End points:

* Proven or probable invasive fungal infection.
* Initiation of full dose parental antifungal therapy for proven or probable invasive fungal infection.
* Successful recovery of ANC more than 1000/cumm or completion of induction.

Study protocol:

* After signing informed consent forms patients will be randomly assigned to a regimen of oral Voriconazole or IV low dose Amphotericin B.
* Oral Voriconazole will be given in dose of 6mg/kg 12 hourly on day1 then 4mg/kg 12 hourly daily or IV Amphotericin B 0.5 mg/kg/day weekly thrice.
* Patient will be started at the time of initiation of induction till completion of induction.

Evaluation:

- Patients will be evaluated at baseline, twice weekly for duration of study and at completion of study.

Baseline evaluation:

* History and physical examination.
* Hemogram and biochemistry
* Chest X ray

Evaluation of patients with baseline fever:

For the patient presenting with fever at baseline (randomization), blood and urine culture for fungus and bacteria will be send, X- ray chest to rule out consolidation at baseline will be done in all patients. The patients will be started on antibiotics as per the routine institutional policy. If patient becomes afebrile before day 5, then antibiotics will be continued for 5 days after becoming afebrile. If patient is still febrile at day 5, then empiric therapeutic antifungal therapy will be added.

Evaluation of patients with breakthrough fever:

In case of patient developing fever >38 degree C (axillary) during induction chemotherapy, patient will be evaluated by clinical examination, hemogram ,biochemistry, chest X ray, blood and urine culture for fungus and bacterial for three consecutive days. Patients with evidence of chest infection on chest X ray/signs and symptoms of chest infection/febrile even after receiving 5 days of appropriate antibiotics will be subjected to HRCT scan of chest. Patients showing consolidation , or signs of chest infection on chest CT will be subjected for broncoscopy and bronchoalveolar lavage. The brochoalveolar lavage will be sent for microscopy (gram staining), culture for fungal and bacterial growth. Full dose therapeutic antifungal will be started earlier in case of development of pneumonia, hemodynamic instability even if before 5 days of antibiotics which will be considered as failure of prophylaxis. Whenever feasible (not mandatory) depending on the patient's clinical condition, we will try to obtain tissue sample for histology by FNAC/Biopsy from the suspected infected site.

ELIGIBILITY:
Inclusion Criteria:

* Patients age </= 15 years with de novo acute leukemia (AML, ALL) undergoing induction chemotherapy.
* No evidence of fungal infection at randomization
* No pneumonia at presentation on CXR.
* No systemic antifungal therapy within 7 days before randomization.

Febrile patients with no pneumonia, systemic fungal infection and hemodynamically stable will be eligible for study.

Exclusion Criteria:

* Patients with baseline pneumonia on CXR.
* Laboratory evidence of significant hepatic or renal dysfunction (defined as a SGOT or SGPT >5 times, Total bilirubin>2 times and Serum creatinine > 2 times upper limit of normal)

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Prevention of possible, probable or proven fungal infection. | Completion of Induction Chemotherapy or successful recovery of ANC > 1000/mm3

CONTACTS AND LOCATIONS:
Overall Officials: SAMEER BAKHSHI, MD, Principal Investigator — Institute Rotary Cancer Hospital, All India Institute of Medical Sciences
Locations (1):
- Institute Rotary Cancer Hospital, All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Mandhaniya S, Iqbal S, Sharawat SK, Xess I, Bakhshi S. Diagnosis of invasive fungal infections using real-time PCR assay in paediatric acute leukaemia induction. Mycoses. 2012 Jul;55(4):372-9. doi: 10.1111/j.1439-0507.2011.02157.x. Epub 2012 Mar 16. PMID 22420668
- [Derived] Mandhaniya S, Swaroop C, Thulkar S, Vishnubhatla S, Kabra SK, Xess I, Bakhshi S. Oral voriconazole versus intravenous low dose amphotericin B for primary antifungal prophylaxis in pediatric acute leukemia induction: a prospective, randomized, clinical study. J Pediatr Hematol Oncol. 2011 Dec;33(8):e333-41. doi: 10.1097/MPH.0b013e3182331bc7. PMID 22042283